CLINICAL TRIAL: NCT05609552
Title: Biodistribution and Pharmacokinetics of Pretomanid in Tuberculosis Patients Using 18F-Pretomanid PET
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00303845; R01HL131829 (NIH)
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Tuberculosis
Keywords: PET/CT; Pretomanid
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tuberculosis patients: Patients with confirmed TB [culture confirmed or positive by genotypic testing with GeneXpert, Accuporobe, etc.] by genotype and/or culture testing positive for M. tuberculosis
  Interventions: Combination Product: 18F-Pretomanid PET/CT

INTERVENTIONS:
Combination Product: 18F-Pretomanid PET/CT — A bolus of less than or equal to 10 mCi (370 MBq) of 18F-pretomanid will be injected into the intravenous line by slow IV push. Immediately after administration of 18F-pretomanid, dynamic PET acquisition will take place.

SUMMARY:
This is an observational study that will examine the pretomanid pharmacokinetics (PK) in tuberculosis (TB) patients. Dynamic 18F-pretomanid PET/CT will be performed after intravenous injection of 18F-pretomanid to determine multi-compartment, noninvasive determination of pretomanid PK in TB patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age at the time of consent and imaging
2. Healthy subjects OR Subjects with confirmed tuberculosis OR high suspicion of active tuberculosis by treating physician.
3. For TB patients: Imaging evidence of suspected tuberculosis infection involving the lung, and possible additional other sites of involvement.
4. For TB patients: After TB diagnosis is confirmed, patients will be eligible to participate up to 6 weeks after starting TB treatment.
5. Subject is willing to give written informed consent. Subject is willing and able to comply with the protocol for the duration of the study including undergoing scheduled visits and study procedures.
6. Screening clinical laboratory values must be within normal limits or judged not clinically significant by the investigator.
7. Women of child-bearing potential (WOCBP) must have a negative serum or urine pregnancy test within 24 hours prior to the radiotracer administration.
8. Patients or their legal representatives must have the ability to read, understand and provide written informed consent for the initiation of any study-related procedures.

Exclusion Criteria:

1. Inadequate venous access
2. Any medical condition that in the judgment of the investigator would make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and female members of all races and ethnic groups are eligible for this trial and encouraged to participate. Subjects from different groups will be enrolled concurrently.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Biodistribution of 18F-pretomanid | Up to 4 hours
  Exposures in infected sites (pneumonia, cavitary lesions, etc.) will compared with the uninfected compartments. Standard units such as area under the curve (AUC) or AUC ratios will be utilized.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay K Jain, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No